CLINICAL TRIAL: NCT00795223
Title: Comparative Effect of 0.2 or 0.3 Spinal Morphine and 0.25 or 0.5 % Bupivacaine for Femoral Nerve Block After Total Knee Replacement
Brief Title: Comparative Pain Control Between 0.2 or 0.3 Spinal Morphine and 0.25 or 0.5 % Bupivacaine for FNB After TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Thitima Chinachoti, Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 461/2551(EC1); Grant by the siriraj Hospital
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Post Operative Pain; Total Knee Replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Injection of 0.3 mg morphine with spinal block and perform femoral nerve block with 0.5% bupivacaine
  Interventions: Drug: morphine and bupivacaine
- 2 (Active Comparator): Injection of 0.3 mg morphine with spinal block and perform femoral nerve block with 0.25% bupivacaine
  Interventions: Drug: spinal morphine and marcaine
- 3 (Active Comparator): Injection of 0.2 mg morphine with spinal block and perform femoral nerve block with 0.5% bupivacaine
  Interventions: Drug: morphine and bupivacaine
- 4 (Active Comparator): Injection of 0.2 mg morphine with spinal block and perform femoral nerve block with 0.25% bupivacaine
  Interventions: Drug: morphine and bupivacaine

INTERVENTIONS:
Drug: morphine and bupivacaine — 0.3 mg morphine for spinal together with 0.5% bupivacaine for femoral nerve block
  Other Names: marcaine
  Arms: 1
Drug: spinal morphine and marcaine — 0.3 mg spinal morphine together with 0.25% bupivacaine for femoral nerve block
  Other Names: marcaine
  Arms: 2
Drug: morphine and bupivacaine — 0.2 mg morphine for spinal 0.5% bupivacaine for femoral nerve block
  Other Names: marcaine
  Arms: 3
Drug: morphine and bupivacaine — 0.2 mg morphine for spinal together with 0.25% bupivacaine for femoral nerve block
  Other Names: marcaine
  Arms: 4

SUMMARY:
Comparative efficacy of 24 and 48 hours post operative pain control in single total knee replacement between intrathecal bupivacaine with 0.2 or 0.3 mg morphine together with 0.25 or 0.5 % bupivacaine for single femoral nerve block

ELIGIBILITY:
Inclusion Criteria:

* Single elective total knee replacement in ASA 1-3 without significant cardiovascular limitation

Exclusion Criteria:

* patient at risk in usage COX-2 for post operative pain control

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Global assessment in post operative pain control | Begining of first enrollment in december 2008

SECONDARY OUTCOMES:
Global assessment of post operative pain in 48 HOURS AND SIDE EFFECTS | first enrollment in December 2008

CONTACTS AND LOCATIONS:
Overall Officials: Thitima Chinachoti, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Bangkoknoi, Thailand